CLINICAL TRIAL: NCT05300139
Title: Validation of Ultrasonic Positive Diagnosis Criteria of Ipsilateral Deep Vein Thrombosis Recurrence of the Lower Limbs Based on Thrombosis Evolution at a 3-month Follow-up Under Anticoagulation: The ULTREC Project Ancillary Study
Brief Title: Ancillary Study of the ULTREC Project
Acronym: ULTRECAncillar
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Intercommunal de Toulon La Seyne sur Mer (Other)
Responsible Party: Sponsor
Other Study IDs: 2021-CHITS-014
Record Dates: First submitted 2022-03-03; First posted 2022-03-29 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Deep Vein Thrombosis
Keywords: Deep vein thrombosis; Recurrence; Colour doppler ultrasound; Diagnostic strategy; Outcome
MeSH Terms: conditions — Venous Thrombosis; Recurrence

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients included in the ULTREC study who had a recurrence of deep vein thrombosis: Patients who have a baseline CDUS diagnosis of recurrent DVT as identified in the ULTREC study.
  Interventions: Other: Color Doppler Ultrasound

INTERVENTIONS:
Other: Color Doppler Ultrasound — Comparison between D90±5 and baseline CDUS
  Other Names: Diagnosis strategy

SUMMARY:
The ULTREC research project is designed to assess the safety of a negative strategy relying on Colour Doppler Ultrasound (CDUS) for excluding the diagnosis of a new thrombosis. The ULTREC project does not take into account the validity of the CDUS positive criteria used to confirm the diagnosis of Deep Vein Thrombosis (DVT) recurrence.

The risk of considering only the negative strategy is to ignore the possibility of having an improvement in sensitivity and negative predictive value at the expense of specificity and positive predictive value and therefore to increase the false positive rate leading to an overdiagnosis of recurrence and an overtreatment, and a potential bleeding risk.

In the ULTREC-ANCILLARY study, the research will aim at assessing the validity of baseline CDUS positive criteria for the diagnosis of DVT recurrence. As there is no diagnostic standard to which the results could be compared, it is suggested to validate these criteria based on the evolution of the thrombosis on CDUS performed at D90±5.

The hypothesis is that an unchanged appearance under anticoagulation would be in favor of sequelae and will invalidate the initial diagnosis (diagnostic failure)

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Known history of objectively documented deep vein thrombosis of the lower limb (with or without pulmonary embolism)
3. Out-patients referred for clinically suspected acute recurrent ipsilateral DVT of the lower limb
4. Patients covered by social security or an equivalent regimen
5. No objection to the use of the data
6. Inclusion in the ULTREC study

Exclusion Criteria:

1. Known current pregnancy
2. Any condition, which may prevent from performing the colour doppler ultrasound test
3. Delay from onset of symptoms to inclusion of more than 10 days
4. Therapeutic anticoagulation for more than 48 hours in the two days prior to consent to ULTREC Study
5. Presence of clinical symptoms or signs of pulmonary embolism
6. Life expectancy less than 3 months
7. Patient unable to adhere to ULTREC protocol follow-up
8. Participants under judicial protection or incapacity

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients included in the ULTREC study who had a recurrence of deep vein thrombosis
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2021-11-29 (Actual); Primary Completion 2023-01-24 (Actual); Study Completion 2023-01-24 (Actual)

PRIMARY OUTCOMES:
Evolution of the thrombosis at D90±5 | 90 days
  Failure rate judged on the stable aspect of the thrombosis at D90±5 defined by the absence of change in the obstruction and the extent of the thrombosis and the absence of change in the venous diameter under compression (no increase or increase < 4 mm). Vein diameter is measured under compression by ultrasound in a cross-sectional view from the external wall to the external wall of the vein segment.

SECONDARY OUTCOMES:
Validation of positive DVT criteria by comparison between D30±2 and baseline CDUS | 30 days
  Failure rate judged on the stable aspect of the thrombosis at D30±2 defined by the absence of change in the obstruction and the extent of the thrombosis and the absence of change in the venous diameter under compression (no increase or increase < 4 mm)
Clinical and Imaging characteristics | 90 days
  Comparison of clinical and CDUS imaging characteristics between day-0 and day-90 visits
Evolution during follow-up | 90 days
  Rate of worsening, stabilization and improvement (regression, normalization) Worsening is defined by : a transition from partial obstruction to complete occlusion of a vein segment, an increase ≥ 4 mm in vein diameter measurement or progression of thrombus to another vein segment.
  Stabilization is defined by : an unchanged pattern. Improvement (regression, normalization) is defined by : a transition from a complete occlusion to a partial obstruction or normalization of the vein segment.
Baseline characteristics for favorable outcome | 1 day
  Imaging and clinical characteristics of thrombus at Day-0 visit
Venous diameter | 90 days
  Evolution of venous diameter at day-90 as measured under compression by ultrasound in a cross-sectional view from the external wall to the external wall of the vein segment
Diagnosis of individual characteristics of DVT recurrence | 90 days
  Failure rate related to the baseline measurement of vein diameter and ULTREC diagnostic recurrence positivity criteria (defined as an occlusive thrombus or a partially obstructive thrombus without reflux, or a free-floating thrombus).

CONTACTS AND LOCATIONS:
Overall Officials: Antoine ELIAS, MD, Study Director — Centre Hospitalier Intercommunal Toulon La Seyne sur Mer
Locations (12):
- France (12):
  - Cabinet d'angiologie Cazanave, Carcassonne, Aude
  - Centre Hospitalier de Carcassonne, Carcassonne, Aude
  - Cabinet d'angiologie Dias, Martigues, Bouches Du Rhône
  - Cabinet d'angiologie De Mari, Ajaccio, Corse-du-Sud
  - Cabinet d'angiologie Secondi, Ajaccio, Corse-du-Sud
  - Cabinet d'angiologie Cazaux, Auch, Gers
  - Centre Hospitalier d'Auch, Auch, Gers
  - Cabinet d'angiologie Bonavita, Bastia, Haute-Corse
  - Clinique Rive Gauche, Toulouse, Haute-Garonne
  - Clinique des fleurs, Ollioules, Var
  - Cabinet d'angiologie Bensedrine, Six-Fours-les-Plages, Var
  - Centre Hospitalier Intercommunal Toulon La Seyne sur Mer, Toulon, Var

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ageno W, Squizzato A, Wells PS, Buller HR, Johnson G. The diagnosis of symptomatic recurrent pulmonary embolism and deep vein thrombosis: guidance from the SSC of the ISTH. J Thromb Haemost. 2013 Aug;11(8):1597-602. doi: 10.1111/jth.12301. No abstract available. PMID 23682905
- [Background] Aguilar C, del Villar V. Combined D-dimer and clinical probability are useful for exclusion of recurrent deep venous thrombosis. Am J Hematol. 2007 Jan;82(1):41-4. doi: 10.1002/ajh.20754. PMID 16947316
- [Background] Bates SM, Jaeschke R, Stevens SM, Goodacre S, Wells PS, Stevenson MD, Kearon C, Schunemann HJ, Crowther M, Pauker SG, Makdissi R, Guyatt GH. Diagnosis of DVT: Antithrombotic Therapy and Prevention of Thrombosis, 9th ed: American College of Chest Physicians Evidence-Based Clinical Practice Guidelines. Chest. 2012 Feb;141(2 Suppl):e351S-e418S. doi: 10.1378/chest.11-2299. PMID 22315267
- [Background] Fraser DG, Moody AR, Morgan PS, Martel AL, Davidson I. Diagnosis of lower-limb deep venous thrombosis: a prospective blinded study of magnetic resonance direct thrombus imaging. Ann Intern Med. 2002 Jan 15;136(2):89-98. doi: 10.7326/0003-4819-136-2-200201150-00006. PMID 11790060
- [Background] Geersing GJ, Zuithoff NP, Kearon C, Anderson DR, Ten Cate-Hoek AJ, Elf JL, Bates SM, Hoes AW, Kraaijenhagen RA, Oudega R, Schutgens RE, Stevens SM, Woller SC, Wells PS, Moons KG. Exclusion of deep vein thrombosis using the Wells rule in clinically important subgroups: individual patient data meta-analysis. BMJ. 2014 Mar 10;348:g1340. doi: 10.1136/bmj.g1340. PMID 24615063